CLINICAL TRIAL: NCT03900299
Title: Tailoring Surgical Management of Multifocal Breast Cancer:is There a Possibility
Brief Title: Evaluating New Surgical Technique in Management of Female Patients With Operable Multifocal Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, mostafa mohamed elsayed, registrar of surgical oncology and general surgery, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: multifocal breast cancer2018
Record Dates: First submitted 2019-03-20; First posted 2019-04-03 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: breast conservative surgery; oncoplastic breast surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All operable(don't require neoadjuvant therapy or inflammatory carcinoma) female patients diagnosed as multifocal breast cancer will receive oncoplastic breast surgery as a surgical treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oncoplastic breast surgery (Other)
  Interventions: Procedure: oncoplastic breast surgery

INTERVENTIONS:
Procedure: oncoplastic breast surgery — oncoplastic breast surgery with level 1 or 2 according to the case using intra operative frozen section to assess the margin

SUMMARY:
Multi-focal Breast Cancers(MFBC) still have undiscoverable Clinical Significance reflecting on a debatable surgical decision for this Category of breast cancer. A prospective study was conducted using certain surgical technique as a surgical treatment for female patients with operable breast cancer managed at the Surgical Oncology Unit, Alexandria University from May. 2017 to May2018 and will be followed for 3 Years.Analysis will be done to settle a paradigm for surgical management of Multi-focal Breast Cancer

DETAILED DESCRIPTION:
* Age at diagnosis: young patients are defined as younger than 35 years.
* Surgical techniques: Preoperatively all patients will undergo physical examination of both breasts and axillae as well as bilateral mammograms and ultrasonography of both breasts. Histopathological diagnosis of cancer will be made prior to surgery. The planned procedure will be discussed. Different oncoplastic techniques will be utilized to achieve oncologically appropriate margins with either sentinel lymph node detection or axillary lymph node dissection according to the triple assessment of the patients . Surgical margins were determined by macroscopic and histologic examination of frozen sections of the breast specimens in the operating room. An adequate safety margin of 1cm was always insured. Breast remodeling will be done according to breast size, degree of ptosis and size of defect.
* Tumor characteristics: size, nodal status, presence of lympho-vascular invasion, amount of intraductal component, tumor grade, margin status, hormone receptor, and Her2 neu status.
* Margins will be regarded as negative when permanent histological examination found no ink on the tumor.
* Postoperative surgical complications will be documented if happened; seroma formation, hematoma and or wound dehiscence.
* Cosmetic outcome: The postoperative esthetic result will be evaluated asking the patients to rate the postoperative cosmetic result and their degree of satisfaction compared to the preoperative breast using a five-point scale (excellent, 5; good, 4; fair, 3; poor, 2;bad, 1). Objective assessment of the cosmetic result was done by two surgeons, rated on a visual analog scale from 1 (unacceptable result) to 10 (excellent result). Evaluation is based on 5 criteria, namely: breast symmetry, glandular tissue defects, nipple and areola reconstruction, scar quality and/or retraction, and the resultant breast shape. (14)
* The occurrence of loco-regional recurrence or distant metastases during the follow-up period was recorded and considered as an end point for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* all operable female patients affected with multifocal breast cancer

Exclusion Criteria:

* inflammatory breast cancer
* patients need receiving neoadjuvant therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — all operable female patients affected with multifocal breast cancer
Enrollment: 114 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2020-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T. Awad, MD, Study Director — professor of surgical oncology,Alexandria university; Mostafa M. Elsayed, Msc, Principal Investigator — Surgical oncology registrar,Alexandria university
Locations (1):
- Faculty of medicine ,Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: will be available for 1 year after publication
Access Criteria: individual participant data will be available to every researcher in field of multi -focal breast cancer, the candidate should have an accepted protocol from the ethical committee of the organization. contacting the main investigator will be method to review the request
URL: http://www.med.alexu.edu.eg/ethics-committee/

REFERENCES:
- [Result] Yerushalmi R, Kennecke H, Woods R, Olivotto IA, Speers C, Gelmon KA. Does multicentric/multifocal breast cancer differ from unifocal breast cancer? An analysis of survival and contralateral breast cancer incidence. Breast Cancer Res Treat. 2009 Sep;117(2):365-70. doi: 10.1007/s10549-008-0265-1. Epub 2008 Dec 11. PMID 19082705
- [Result] Gentilini O, Botteri E, Rotmensz N, Da Lima L, Caliskan M, Garcia-Etienne CA, Sosnovskikh I, Intra M, Mazzarol G, Musmeci S, Veronesi P, Galimberti V, Luini A, Viale G, Goldhirsch A, Veronesi U. Conservative surgery in patients with multifocal/multicentric breast cancer. Breast Cancer Res Treat. 2009 Feb;113(3):577-83. doi: 10.1007/s10549-008-9959-7. Epub 2008 Mar 11. PMID 18330695
- Available data/document: Study Protocol — http://www.med.alexu.edu.eg/ethics-committee/

RESULTS

PARTICIPANT FLOW:
Groups:
- Multifocal Breast Cancer Patients Treated Surgically by MRM: multifocal breast cancer patients involved in the study will be randomized to be treated either by oncoplastic breast conserving surgery or modified radical mastectomy(MRM)
- Multifocal Breast Cancer Patients Treated Surgically by OPS: multifocal breast cancer patients involved in the study randomized in the setting of receiving surgical treatment either modified radical mastectomy (MRM) or oncoplastic breast surgery(OPS)
Period: Overall Study
Arm/Group | Multifocal Breast Cancer Patients Treated Surgically by MRM | Multifocal Breast Cancer Patients Treated Surgically by OPS
Started | 56 | 58
Completed | 56 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multifocal Breast Cancer Patients Treated Surgically by MRM | Multifocal Breast Cancer Patients Treated Surgically by OPS | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Customized [Count of Participants; unit: Participants] — Age in years
  < 40 40- 50- 60+
  Participants
    <40 | 3 | 5 | 8
    40-49 | 10 | 18 | 28
    50-59 | 14 | 14 | 28
    60+ | 29 | 21 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 58 | 114
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 56 | 58 | 114
tumor size [Count of Participants; unit: Participants] — T(TUMOR SIZE) T1 <2 cm T2 (2-5 cm) T3 > 5 cm T4 tumor attached to the skin
  Participants
    T1 | 23 | 34 | 57
    T2 | 32 | 24 | 56
    T3 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of the Tumor
Description: assessment of the occurrence of local or distant recurrence through:
  1. monthly clinical examination of both breast and axillae
  2. monthly liver functions tests and complete blood count
  3. radiological assessment if clinically indicated
Time Frame: a median of 30 months post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Multifocal Breast Cancer Patients Treated Surgically by MRM | Multifocal Breast Cancer Patients Treated Surgically by OPS
Number analyzed (Participants) | 56 | 58
Participants
  Tumor recurrence | 2 | 3
  no tumor recurrence | 54 | 55

2. Secondary Outcome: Cosmetic Result
Description: assessment of breast cosmesis after oncoplastic surgical intervention.Evaluation is based on 5 criteria, namely: breast symmetry, glandular tissue defects, nipple and areola reconstruction, scar quality and/or retraction, and the resultant breast shape.
  each criteria will be evaluated either satisfactory or not,satisfactory evaluation will represent 1 point.
  unsatisfactory will represent 0 point excellent result is equal or more than 4 points good result is equal to 3 points fair result is equal to 2 points bad result is equal to 1 point or less
Time Frame: a median of 30 months post operative
Population: overall number of participants subjected to oncoplastic breast surgery is 58 subdivided to categories according to the oncoplastic technique used, totally 58 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Oncoplastic Breast Surgery
Number analyzed (Participants) | 58
Participants
  theraputic lateral mammoplasty: number analyzed (Participants) | 20
  theraputic lateral mammoplasty: excellent cosmetic result | 13
  theraputic lateral mammoplasty: very good cosmetic result | 7
  round block: number analyzed (Participants) | 14
  round block: excellent cosmetic result | 13
  round block: very good cosmetic result | 1
  parallelogram mastopxy: number analyzed (Participants) | 9
  parallelogram mastopxy: excellent cosmetic result | 7
  parallelogram mastopxy: very good cosmetic result | 2
  V theraputic mammoplasty: number analyzed (Participants) | 4
  V theraputic mammoplasty: excellent cosmetic result | 3
  V theraputic mammoplasty: very good cosmetic result | 1
  Latissimus Dorsi flap: number analyzed (Participants) | 3
  Latissimus Dorsi flap: excellent cosmetic result | 1
  Latissimus Dorsi flap: very good cosmetic result | 2
  J theraputic mammoplasty: number analyzed (Participants) | 4
  J theraputic mammoplasty: excellent cosmetic result | 3
  J theraputic mammoplasty: very good cosmetic result | 1
  grisotti flap: number analyzed (Participants) | 2
  grisotti flap: excellent cosmetic result | 1
  grisotti flap: very good cosmetic result | 1
  reduction therapeutic mammoplasty: number analyzed (Participants) | 2
  reduction therapeutic mammoplasty: excellent cosmetic result | 1
  reduction therapeutic mammoplasty: very good cosmetic result | 1

ADVERSE EVENTS:
Time Frame: through 24 months post operative
Description: Early complications
  1. Haematoma
  2. Seroma
  3. Abcess
  4. Skin or NAC necrosis
  Late complications
  1. Scar fibrosis
  2. keloid
  3. steatonecrosis
Groups:
- Multifocal Breast Cancer Patients Treated Surgically by MRM: multifocal breast cancer patient treated by modified radical mastectomy(MRM) 66 patients
  Early complications Haematoma 2 patients out of 56 Seroma 16 patients out of 56 Skin or flap necrosis 5 patients out of 56 Abcess 3 patients out of 56
  Late complications Scar fibrosis 2 patients out of 56 keloid 1 patients out of 56
- Multifocal Breast Cancer Patients Treated Surgically by OPS: multifocal breast cancer patients treated by oncoplastic breast surgery(OPS) 58 patients
  Early complications Haematoma 2 patients out of 58 Seroma 10 patients out of 58 Abcess 4 patients out of 58 Skin or NAC necrosis 2 patients out of 58
  Late complications Scar fibrosis 3 patients out of 58 keloid 2 patients out of 58 steatonecrosis 5 patients out of 58
Arm/Group | Multifocal Breast Cancer Patients Treated Surgically by MRM | Multifocal Breast Cancer Patients Treated Surgically by OPS
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 29/56 | 28/58
Other Adverse Events (participants affected / at risk) | 0/56 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multifocal Breast Cancer Patients Treated Surgically by MRM (N=56) | Multifocal Breast Cancer Patients Treated Surgically by OPS (N=58)
Haematoma (Surgical and medical procedures) | 2 (2) | 2 (2) — Early post operative complication
Seroma (Surgical and medical procedures) | 16 (16) | 10 (10) — Early post operative complications
skin necrosis (Surgical and medical procedures) | 5 (5) | 2 (2) — Early post operative complications
abcess (Surgical and medical procedures) | 3 (3) | 4 (5) — early post operative
Scar fibrosis (Surgical and medical procedures) | 2 (2) | 3 (3) — Late post operative complications
keloid (Surgical and medical procedures) | 1 (1) | 2 (2) — late post operative complications
steatonecrosis (Surgical and medical procedures) | 0 (0) | 5 (5) — late post operative complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03900299/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03900299/SAP_001.pdf